CLINICAL TRIAL: NCT04401618
Title: Retrospective Clinical Evaluation of RMGI/GI Class V Restorations Placed by Dental Students
Brief Title: Retrospective Evaluation of RMGI/GI Class V Restorations
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Maria Jacinta Santos, Associate Professor, Western University, Canada
Other Study IDs: 107864
Record Dates: First submitted 2020-05-14; First posted 2020-05-26 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Material, Dental
Keywords: Glass-Ionomer Cement; Polyacid-Modified Composite Resin; Dental School

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Class V RMGI Restorations: Resin-modified glass ionomer (RMGI - Fuji 2 LC) Class V restorations performed by by 3rd and 4th-year dental students in adult patients of Schulich dental clinic over the last three years will be evaluated using mirrors and probes.
  Interventions: Other: Retrospective evaluation of RMGI and GIC Class V Restorations
- Class V Glass ionomer - GIC Restorations: Glass ionomer (GI - Fuji 9) Class V restorations performed by by 3rd and 4th-year dental students in adult patients of Schulich dental clinic over the last three years will be evaluated using mirrors and probes.
  Interventions: Other: Retrospective evaluation of RMGI and GIC Class V Restorations

INTERVENTIONS:
Other: Retrospective evaluation of RMGI and GIC Class V Restorations — Retrospective evaluation of RMGI and GIC Class V Restorations that were placed by dental students over the last three years were evaluated using the modified USPHS criteria using mirrors and probes.

SUMMARY:
Brief Summary: Retrospective study to evaluate the clinical performance of two restorative materials - glass-ionomer (GI) and resin-modified glass-ionomer (RMGI) materials - in Class V carious and non-carious cervical lesions restored by dental students.

DETAILED DESCRIPTION:
The aim of this retrospective study was to evaluate the clinical performance of glass-ionomer (GI) and resin-modified glass-ionomer (RMGI) materials in Class V carious and non-carious cervical lesions restored by dental students. Ninety-six (96) restorations performed with either GI (Fuji IX) (n=39) or RMGI (Fuji II) (n=57) were evaluated using the modified USPHS (United States Public Health Systems) criteria by two independent investigators at two follow-up evaluations (two years apart). The Fisher statistical test was used to compare USPHS criteria and examine significant differences by setting p<0.05 for statistical significance and the Kaplan-Meier algorithm was used to calculate the survival probability.

ELIGIBILITY:
Inclusion Criteria:

• Class V Ionomer restorations (RMGI and GIC) placed by 3rd and 4th dental students over the last three years.

Exclusion Criteria:

* Class V Restorations placed outside of the dental school
* Class V Restorations that used other restorative materials Class V Ionomer restorations (RMGI and GIC0 placed before three years on the time of evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults that have Class V Ionomer restorations (RMGI and GIC) placed by 3rd and 4th dental students at the Schulich Dental Clinic over the last three years.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Post-Operative Sensitivity | 2 years
  Absence of sensitivity to pressure, cold or hot temperature on the teeth restored (checked verbally by inquiring the patient about the presence or absence of pain in the presence of stimuli)
Secondary Caries | 2 years
  No visual evidence of dark, deep discolouration or cavitation adjacent to the restoration (visually and manually checked with the tip of a dental hand instrument - explorer)
Anatomic Form | 2 years
  Restoration's anatomy is continuous with existing anatomic form of remaining tooth structure (checked visually with a dental intra-oral mirror)
Color match | 2 years
  No difference between the tooth and restoration colour (checked visually with a dental intra-oral mirror)
Surface Roughness | 2 years
  Surface texture of the restoration is similar to tooth structure (manually checked with the tip of a dental hand instrument - explorer)
Marginal Discolouration | 2 years
  No visual evidence of dark discolouration adjacent to the margins of the restoration (checked visually with a dental intra-oral mirror)
Marginal Integrity | 2 years
  Restoration closely adapted to the tooth. No crevice visible (manually checked with the tip of a dental hand instrument - explorer)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jacinta Santos, Ph.D, Principal Investigator — Schulich Dentistry-Western University
Locations (1):
- Schulich Medicine and Dentistry - Western University, London, Ontario, Canada

REFERENCES:
- [Background] Santos MJ, Ari N, Steele S, Costella J, Banting D. Retention of tooth-colored restorations in non-carious cervical lesions--a systematic review. Clin Oral Investig. 2014;18(5):1369-81. doi: 10.1007/s00784-014-1220-7. Epub 2014 Mar 27. PMID 24671713
- [Background] Neo J, Chew CL, Yap A, Sidhu S. Clinical evaluation of tooth-colored materials in cervical lesions. Am J Dent. 1996 Feb;9(1):15-8. PMID 9002808
- [Background] Franco EB, Benetti AR, Ishikiriama SK, Santiago SL, Lauris JR, Jorge MF, Navarro MF. 5-year clinical performance of resin composite versus resin modified glass ionomer restorative system in non-carious cervical lesions. Oper Dent. 2006 Jul-Aug;31(4):403-8. doi: 10.2341/05-87. PMID 16924979
- [Background] van Dijken JW. Retention of a resin-modified glass ionomer adhesive in non-carious cervical lesions. A 6-year follow-up. J Dent. 2005 Aug;33(7):541-7. doi: 10.1016/j.jdent.2004.11.015. Epub 2005 Feb 8. PMID 16005793
- [Background] Imbery TA, Namboodiri A, Duncan A, Amos R, Best AM, Moon PC. Evaluating dentin surface treatments for resin-modified glass ionomer restorative materials. Oper Dent. 2013 Jul-Aug;38(4):429-38. doi: 10.2341/12-162-L. Epub 2012 Oct 22. PMID 23088188